CLINICAL TRIAL: NCT01049490
Title: Safety and Efficacy of Dose Sparing Intradermal S-OIV H1N1 Influenza Vaccination With the Novel Microneedle Delivery Device
Brief Title: Dose Sparing Intradermal S-OIV H1N1 Influenza Vaccination Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr Ivan FN Hung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HKU-2009-128
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Influenza Infection
Keywords: Intradermal vaccination, H1N1, microneedle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramuscular (Active Comparator): 15 mcg H1N1 vaccine delivered via intramuscular injection (control)
  Interventions: Biological: S-OIV H1N1 vaccine
- Intradermal (Active Comparator): Intradermal: H1N1 vaccine delivered via intradermal injection: Experimental
  Interventions: Biological: S-OIV H1N1 vaccine

INTERVENTIONS:
Biological: S-OIV H1N1 vaccine — Intramuscular: 15 mcg H1N1 vaccine: Control Intradermal: 3 mcg S-OIV H1N1 vaccine: Interventional

SUMMARY:
Primary objective: To evaluate the safety and immunogenicity of low-dose ID S-OIV H1N1 vaccines delivered via a novel microneedle device (MicronJet600) and compare this to the full-dose standard IM injection.

Hypothesis: Low dose (20%) intradermal (ID) S-OIV H1N1 vaccine delivered via a novel microneedle device (MicronJet600) is equally effective as full-dose standard intramuscular (IM) vaccine.

DETAILED DESCRIPTION:
This is a prospective randomised, single-blinded trial in Queen Mary Hospital. We aim to recruit 200 subjects [with a minimum of 80 subjects per age group (21-65 with chronic diseases and age 65+)] who would be qualified for the Hospital Authority (HA)/ Centre for Health Protection (CHP) Mass Vaccination Program for S-OIV H1N1. These patients include all elderly at the age of 65 or above and all adult patients at the age of 21 or above with chronic illness. Subjects will be randomly assigned to receive either the full-dose (1 dose) standard Panenza vaccine at day 0 (15ug non-adjuvanted monovalent influenza A(H1N1) 2009 vaccine) delivered intramuscularly using a conventional needle (IM group) or a low-dose (1 dose) intradermal injection of Panenza vaccine at day 0 (3ug non-adjuvanted monovalent influenza A(H1N1) 2009 vaccine) delivered with the MicronJet600 (ID group).

ELIGIBILITY:
Inclusion Criteria:

* All participants qualified for the HA/ CHP Mass Vaccination Program for S-OIV H1N1 as stated above: including all elderly at the age of 65 or above and all adult patients at the age of 21 or above with chronic illness including hypertension, diabetes mellitus, ischemic heart disease, cerebrovascular disease, thyroid disease and chronic renal failure.
* All patients give written informed consent.
* Subjects must be available to complete the study and comply with study procedures.
* Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

* Clinically significant immune-related diseases, significant recent co-morbidities and pregnant volunteers.
* Inability to comprehend and to follow all required study procedures.
* History or any illness that might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
* Have received an S-OIV H1N1 vaccination.
* Have a recent (starting May 2009) history (documented, confirmed or suspected) of a flu-like disease).
* Have a known allergy to eggs or other components of the Study Vaccines (including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein), or history of any anaphylaxis, serious vaccine reactions, to any excipients.
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination, or women who are breastfeeding.
* Female of childbearing potential, not using any acceptable contraceptive methods for at least 2 months prior to study entry or that do not plan to use acceptable birth control.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate on day 21 as measured by S-OIV H1N1 specific neutralizing antibody (NT) and hemagglutination inhibition (HAI) in the intradermal (ID) and intramuscular (IM) groups | Day 21

SECONDARY OUTCOMES:
Seroconversion rate day 42 | Day 21 and 42
Geometric mean titer increases in antibodies | Day 21 and 42
Specific neutralizing antibody (NT) titre | Day 21 and 42
Seroprotection rate | Day 21 and 42
Adverse events (30 minutes post vaccination period) | Day 21 and 42

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD MRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Guangdong, China